CLINICAL TRIAL: NCT03291301
Title: The Efficacy of Cognitive Behavioral Therapy (CBT) and Acupressure for Insomnia: A Pilot Randomized Controlled Trial
Brief Title: Group Cognitive Behavioral Therapy and Acupressure for Insomnia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fiona YY Ho, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PSY001
Record Dates: First submitted 2017-09-15; First posted 2017-09-25 (Actual); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Insomnia
Keywords: Insomnia; Cognitive Behavioral Therapy; CBT-I; Acupressure; Traditional Chinese Medicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy; Acupressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT Group (Experimental): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Combined Group (Experimental): Cognitive Behavioral Therapy for Insomnia plus Acupressure
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia; Other: Acupressure
- Wait-list Control Group (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia including psychoeducation, sleep restriction, stimulus control, cognitive restructuring, and relaxation.
  Arms: CBT Group; Combined Group
Other: Acupressure — Acupressure, a non-invasive therapy, is commonly used in Traditional Chinese Medicine
  Arms: Combined Group

SUMMARY:
This study will examine the use of cognitive behavioural therapy (CBT) and acupressure in treating insomnia in Chinese adults. The main components of CBT for insomnia (CBT-I) includes psychoeducation, sleep restriction, stimulus control, cognitive restructuring, and relaxation. CBT-I is widely used in western countries but it fails to address patient preference among Chinese adults with insomnia, as demonstrated in a previous study examining the subjective experience of chronic insomnia in Hong Kong Chinese adults. The study revealed that Chinese adults showed distrust in hypnotics and preferred traditional Chinese medicine (TCM) which was believed to be more natural. In order to maximize the therapeutic effects of psychological interventions for insomnia, integrative medicine with a combination of CBT-I and TCM could be an alternative to address insomnia in the Chinese population. Acupressure, a non-invasive therapy, is commonly used in TCM. It is suggested that acupressure can induce relaxation and improve sleep quality. Some studies have demonstrated the separate efficacy of CBT-I and acupressure in treating insomnia. However, few studies have examined the effect of their combination.

ELIGIBILITY:
Inclusion Criteria:

1. Hong Kong residents who are able to communicate in Cantonese;
2. Aged ≥ 18 years;
3. A current clinical DSM-5 diagnosis of insomnia disorder according to the Sleep Condition Indicator (SCI) ≥ 21;
4. Insomnia Severity Index (ISI) score ≥ 8; and
5. Willing to give informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Have suicidal ideation based on Beck Depression inventory (BDI-II) Item 9 score ≥ 2 ;
2. Receiving psychotherapy, acupuncture, and/or practitioner-delivered acupressure treatment for insomnia in the past 6 months;
3. Pregnancy; and
4. Taking herbal remedies, over-the-counter medication, or psychotropic drugs that target insomnia within 2 weeks prior to the baseline assessment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change in Insomnia Severity Index | Pre-treatment, 1-week post-treatment and 4-week post treatment
  A 7-item scale designed to evaluate perceived insomnia severity. Ratings on the 5-point Likert scale are obtained on the perceived severity of sleep-onset, sleep-maintenance, early morning awakening problems, satisfaction with current sleep pattern, interference with daily functioning, noticeably of impairment attributed to the sleep problem, and level of distress caused by the sleep problem.

SECONDARY OUTCOMES:
Change in 7-Day Sleep Diary | Pre-treatment, 1-week post-treatment and 4-week post treatment
  The standardized sleep diary records sleep-onset latency (SOL; min), wake after sleep onset (WASO; min), total wake time (TWT; min), total sleep time (TST; min), time in bed (TIB; min); sleep efficiency (SE; calculated as TST/TIB * 100%), etc.
Change in Hospital Anxiety and Depression Scale (HADS) | Pre-treatment, 1-week post-treatment and 4-week post treatment
  A 14-item self-rating scale that measures anxiety and depression in both hospital and community settings. It is divided into an Anxiety subscale (HADS-A) and a Depression subscale (HADS-D) both containing seven intermingled items. It is for screening purpose and not meant to be a diagnostic tool.
Change in Dysfunctional Beliefs and Attitudes about Sleep Scale - 16-item version (DBAS-16) | Pre-treatment, 1-week post-treatment and 4-week post treatment
  A 16-item self-report measure designed to evaluate sleep related cognitions (e.g., faulty beliefs and appraisals, unrealistic expectations, perceptual and attention bias).
Change in Multidimensional Fatigue Inventory (MFI) | Pre-treatment, 1-week post-treatment and 4-week post treatment
  A 20-item self-report instrument designed to measure fatigue. Ratings on a 5-point Likert scale are obtained on the dimensions of general fatigue, physical fatigue, mental fatigue, reduced motivation and reduced activity.
Change in Short Form (Six-Dimension) Health Survey - The Chinese (Hong Kong) Version (SF-6D) | Pre-treatment, 1-week post-treatment and 4-week post treatment
  A preference-based single index measure of health. A six-digit number represents each SF-6D health state, each digit denotes the level of one of six SF-6D dimensions: physical functioning, role limitation, social functioning, bodily pain, mental health, and vitality.

OTHER OUTCOMES:
Change in Credibility-Expectancy Questionnaire (CEQ) | Pre-treatment and 1-week post-treatment
  The 6-item CEQ yielded ratings of treatment credibility, acceptability/satisfaction, and expectations for success.

CONTACTS AND LOCATIONS:
Locations (2):
- Hong Kong (2):
  - The Chinese University of Hong Kong, Hong Kong
  - The Chinese University of Hong Kong, Shatin